CLINICAL TRIAL: NCT03576560
Title: Selective Use of Antibiotics in Neonates Born to Mothers With Suspected Chorioamnionitis
Acronym: Chorio
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: 16NE-Z035-6145
Record Dates: First submitted 2018-06-26; First posted 2018-07-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chorioamnionitis
MeSH Terms: conditions — Chorioamnionitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective Chart Review — Retrospective Chart Review

SUMMARY:
Retrospective Chart Review to determine the selective use of antibiotics in neonates born to mothers with suspected chorioamnionitis

DETAILED DESCRIPTION:
To determine the incidence and types of adverse outcomes in infants born to mothers with signs of chorioamnionitis when these infants are asymptomatic and are not treated with antibiotics empirically.

ELIGIBILITY:
Inclusion Criteria:

• Mother/baby dyads in which the mother was diagnosed with chorioamnionitis and/or had intrapartum fever (as diagnosed by obstetrician)

Exclusion Criteria: None

Ages: 35 Weeks to 42 Weeks | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Mother/baby in which the mother was diagnosed with chorioamnionitis and/or had intrapartum fever
Study Population: Patients born at Women's Hospital/Cone Health in Greensboro, NC, from July, 2012 (when EMR was implemented), to present.
Sampling Method: Non-Probability Sample
Enrollment: 768 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Infants born to mother with chorioamnionitis/intrapartum fever as assessed by chart review. | Infants born from July, 2012 to December 31, 2018.
  The retrospective chart review would analyze the total number of infants born to mothers with chorioamnionitis/intrapartum fever.

CONTACTS AND LOCATIONS:
Overall Officials: John Wimmer, MD, Principal Investigator — MEDNAX Employee
Locations (1):
- Women's Hospital of Greensboro, Greensboro, North Carolina, United States